CLINICAL TRIAL: NCT00892424
Title: Phase I/II Trial of Radiation Therapy and Sorafenib for Treatment of Unresectable Liver Metastases
Brief Title: Sorafenib-RT Treatment for Liver Metastasis (SLIM)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 08-0598-C
Record Dates: First submitted 2009-05-01; First posted 2009-05-04 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Liver Metastasis; Cancer
Keywords: Liver metastasis; sorafenib; Liver metastasis from cancer
MeSH Terms: conditions — Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib + RT (Experimental)
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — Sorafenib doses will be 200mg twice daily orally for 28 days in level I, 400 mg in the morning and 200mg in the evening in level II, and 400mg twice daily orally for 28 days in level III . Radiotherapy will be started at day 8, patients will receive a total of 6 fractions over 2 weeks. Patients will be assessed weekly during treatment, 1 month post-tx, then at 3-month intervals for up to a year after tx, and then followed-up at 6-month intervals up to 3 years.

SUMMARY:
Cancers that have spread to the liver from the primary cancer location (liver metastases) that cannot be removed surgically (unresectable) can be treated with chemotherapy and/or radiation therapy. Previous research has shown that tumours often have abnormal blood vessels that may reduce the effect of radiation therapy. New drugs, known as "anti-angiogenic" drugs have been shown in animal and human studies to damage or change tumour blood vessels in ways that may make tumors more sensitive to radiation treatment. 32- 44 Patients diagnosed with unresectable liver metastasis will be invited to take part in this study. The purpose of this study is to investigate the use of a new anti-angiogenic drug called Sorafenib, in combination radiation therapy and chemotherapy. The study will test how effective the new treatment is, the side effects associated with the new treatment, and to help establish safe dosages of the study medication.

DETAILED DESCRIPTION:
In this study, Stereotactic Body Radiation Therapy(SBRT) and Whole Liver Radiotherapy (WLRT) will be used concurrently with sorafenib at 3 different dosages to determine the tolerability and efficacy of this combined treatment. Sorafenib doses will be 200mg twice daily orally for 28 days in level I, 400 mg in the morning and 200mg in the evening in level II, and 400mg twice daily orally for 28 days in level III . Radiotherapy will be started at day 8, patients will receive a total of 6 fractions over 2 weeks. Patients will be assessed weekly during treatment, 1 month post-tx, then at 3-month intervals for up to a year after tx, and then followed-up at 6-month intervals up to 3 years. Once the Maximum Tolerated Dose (MTD) is established, an expanded cohort for each stratum will accrue such that a total of 10 patients per strata. This will allow us to gain further experience with this regimen and consolidate the safety and efficacy data. Quality of Life (QOL) assessment will be carried out at baseline and 1/3/6/9 mos post-tx. Patients will also be offered correlative studies looking at biomarkers through tissue, blood, and urine samples, and an imaging study looking at tissue perfusion.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed liver metastases
* Largest burden of disease should be hepatic if there's extrahepatic disease exists
* Tumour should be medically inoperable
* Patient have a life expectancy of at least 3 months and a KPS performance status of at least 60%.
* Patient should be 18 years of age or older
* Patient should have adequate organ function
* Patient have Creatinine ≤ 2 times upper limit of normal range
* Patient recovered from the effects of prior therapy
* Patient (or person representing the patient) should be able to give informed consent
* Patient have Child's A score (5 or 6) score
* For women of childbearing age, birth control is being used and the pregnancy test is negative

Exclusion Criteria:

* No major surgery in the past 4 weeks.
* No previous use of sorafenib previously.
* Patient should not have or is receiving systemic therapy or investigational agents within 2 weeks of radiotherapy
* No previous upper abdominal radiation therapy to the liver.
* No serious medical conditions that may be aggravated by treatment, including but not limited to: myocardial infarction within 6 months, congestive cardiac failure, unstable angina, active cardiomyopathy, unstable ventricular arrhythmia, uncontrolled hypertension, uncontrolled psychotic disorders,serious infections, active peptic ulcer disease, active liver disease or previous stroke.
* Patients who are infected with human immunodeficiency virus (HIV), should not be receiving combination anti-retroviral therapy
* No clinically significant liver failure (i.e. encephalopathy or ascites found clinically).
* No thrombolytic therapy within 4 weeks or are they receiving other anticoagulant therapy.
* No underlying cirrhosis with Child's B or C score.
* No history of uncontrolled, life threatening malignancy within the past 6 months.
* Patient should not have a variceal bleed or other gastrointestinal bleed in the past 2 months.
* No brain metastases
* Patient should not be pregnant.
* Patients on Rifampin, St. John's Wort, Phenytoin, Carbamazepine, Phenobarbital, or Chronic use (more than 4 weeks) of dexamethasone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2008-11 (Actual); Primary Completion 2020-09-08 (Actual); Study Completion 2020-09-08 (Actual)

PRIMARY OUTCOMES:
Determine the MTD of sorafenib and RT in patients with liver metastases using an iso-toxicity radiation dose allocation scheme. Determine the acute toxicity (< 3 months) of sorafenib when combined with RT in patients with liver metastases. | 2 years enrollment; 3 years follow-up

SECONDARY OUTCOMES:
Document any observed late toxicities of treatment. Determine 1) the in-field local control based on CT response at 3 months;2)the time to progression and overall survival of this cohort, 3)changes in quality of life in these patients | 2 years enrollment; 3 years follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Laura Dawson, MD, Principal Investigator — University Health Centre, Princess Margaret Cancer Centre
Locations (1):
- University Health Network, Toronto, Ontario, Canada